CLINICAL TRIAL: NCT06359548
Title: PEELED INTERNAL LIMITING MEMBRANE REPOSITION FOR IDIOPATHIC MACULAR HOLES: A Single-centre, Randomized, Prospective Controlled Trial
Brief Title: PEELED INTERNAL LIMITING MEMBRANE REPOSITION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XH-24-002
Record Dates: First submitted 2024-03-29; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-01

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reposition Group (Experimental): Peeled ILM Reposition
  Interventions: Procedure: Peeled ILM Reposition
- Peeling Group (Active Comparator): ILM Peeling
  Interventions: Procedure: ILM Peeling

INTERVENTIONS:
Procedure: Peeled ILM Reposition — The ILM was stained using 0.1 mL of indocyanine green（ICG) for approximately 1minute after PPV. The ILM was grasped with end gripping forceps (Grieshaber Maxgrip 723.13; Alcon Laboratories Inc) at a point away from the center of MH around one disc diameter in inferior quadrant of macular area. First, a horizontal ILM strip was peeled off with a width approximately 1.5 to 2.5 disc diameter. Then, the edge of the horizontal ILM strip was grasped and peeled from inferior to superior area continuously.Then the "ILM roll" was flattened back to peeled area assisted with approximately 1.0 mL of PFO (Perfluoron, Alcon Laboratories, Inc). The position of the fixed ILM flap was adjusted under PFO bubble using flute needle or forceps if required.
  Other Names: ILM Flap reposition; ILM Flap covering
  Arms: Reposition Group
Procedure: ILM Peeling — The ILM was stained using 0.1 mL of indocyanine green（ICG) for approximately 1minute after PPV. The ILM was grasped with end gripping forceps (Grieshaber Maxgrip 723.13; Alcon Laboratories Inc). The strand of ILM was peeled off radially from the foveal center to the vascular arcade. As a result, a round-shaped, 2.5-disk diameter to 3.5-disk diameter ILM-peeled area was created.
  Arms: Peeling Group

SUMMARY:
Macular hiatus (MH) refers to a tissue defect in the photoreceptor cell layer of the inner boundary membrane of the optic disc in the macular region. Among them, idiopathic macular hiatus (IMH) is more common in people over 60 years old and is a common eye disease. With the aging of society, the number of patients increases, and it severely damages the patients' vision and life quality. Previously, the conventional surgical approach for treating MH was vitrectomy combined with inner limiting membrane (ILM) peeling. Although the closure rate of MH is high, many damages to the morphology and function of the ILM peeled area have been found. Our team firstly report a novel technique of peeled ILM reposition. Compared to traditional ILM peeling, the novel technique peeled ILM reposition maintains the integrity of internal retina by "pull" back the ILM flap. The previous pilot clinical study suggests that the novel technique peeled ILM reposition surgical intervention can achieve better morphology and functional prognosis. However, there is currently a lack of larger sample size prospective randomized controlled studies to further clarify the clinical efficacy of this new surgical technique in treating IMH. This study aims to conduct a single center, prospective, and randomized controlled study, combined with previous work, to analyze the efficacy of this novel technique peeled ILM peeling in the treatment of IMH. We hypothesize that this novel technique can achieved better morphological and functional prognosis compared to traditional ILM peeling.

ELIGIBILITY:
Inclusion Criteria:

1. The patients are diagnosed as MH with a diameter ≤ 600 µm by optical coherence tomography.
2. Age ranges from 50 to 80 years.
3. Do not participate in other clinical studies.
4. Agree to sign an informed consent form with good compliance.

Exclusion Criteria:

1. Traumatic macular hole.
2. Combined with serious epiretinal membrane.
3. Combined with diabetic retinopathy, hypertensive retinopathy.
4. Combined with other ocular diseases, such as keratitis，uveitis，retinal vasculitis.
5. Spherical equivalent ≥ -6.0 diopters or axial length ≥ 26 mm.
6. History of intraocular surgery.
7. Presence of staphyloma.
8. Other ocular diseases that influence macular microstructure or visual function.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The change in the best corrected visual acuity (BCVA) from baseline to 6 months postoperatively | Pre-operatively, 1-month postoperatively, 3-month postoperatively, 6-month postoperatively,
  The change of BCVA from baseline to 6-month postoperatively

SECONDARY OUTCOMES:
The MH closure rate | 1-month postoperatively
  The MH closure rate at 1-month postoperatively
The range of inner retinal dimpling | 1-month postoperatively, 3-month postoperatively, 6-month postoperatively,
  The range of inner retinal dimpling was measured by OCT (RTVueXR Avanti; Optovue Inc, Fremont, CA)
Postoperative retinal thickness | Pre-operatively, 1-month postoperatively, 3-month postoperatively, 6-month postoperatively,
  With the Thickness Map protocol of the OCT, the full retinal thickness (from ILM to retinal pigment epithelium), inner retinal thickness (from ILM to inner plexiform layer (IPL)), and outer retinal thickness (from IPL to retinal pigment epithelium) of the fovea, parafovea, and perifovea were recorded, respectively.
The fixation stability and sensitivity threshold | Pre-operatively, 3-month postoperatively, 6-month postoperatively,
  Measured by microperimetry (MAIA, CenterVue, Italy)
mfERG P1 wave density amplitudes | Pre-operatively, 3-month postoperatively, 6-month postoperatively,
  Measured by multifocal electroretinogram (mfERG, Espion, Diagnosys LLC, Cambridge, United Kingdom)
M-score values | Pre-operatively, 1-month postoperatively, 3-month postoperatively, 6-month postoperatively,
  Metamorphopsia score (M-score) measurement was performed using the M-chart (Inami Co, Tokyo, Japan)
NEI-VFQ-25 questionnaire scores | Pre-operatively, 1-month postoperatively, 3-month postoperatively, 6-month postoperatively,
  The scores obtain from National Eye Institute 25-Item Visual Function Questionnaire (NEI-VFQ-25 questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Tian Tian, MD，PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiaotong University Medicine School, Shanghai, China